CLINICAL TRIAL: NCT03189225
Title: Capillary And Venous Accuracy: LifeScan Products vs Hospital Reference and YSI
Acronym: CAVALRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3149479
Record Dates: First submitted 2016-09-20; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capillary And Venous Accuracy (Other): All subjects provided blood sample(s) to be tested on three Blood Glucose Monitoring Systems ( OneTouch Ultra 2, OneTouch Verio (Rice), OneTouch SelectPlus), LifeScan reference instrument ( YSI 2300) and hospitals own biochemistry analysers.
  Interventions: Other: Capillary And Venous Accuracy

INTERVENTIONS:
Other: Capillary And Venous Accuracy — Capillary And Venous Accuracy: LifeScan Products vs Hospital Reference instrument and LifeScan reference instrument (YSI 2300)

SUMMARY:
This study is to evaluate accuracy between product platforms in the hands of users, comparing capillary to venous response vs YSI reference instrument as well as the local hospital analyser.

DETAILED DESCRIPTION:
This study will gather data to:

* Determine if extreme bias can be observed between 3 candidate products for user accuracy.
* Assess the offset between venous blood samples versus capillary blood samples.
* Determine if there are measurable donor factors which influence the product bias.
* Assess any offset between YSI 2300 reference instruments and hospital laboratory analyser and impact on bias difference between BGM product types.

ELIGIBILITY:
Summary of Inclusion Criteria:

* Male or Female subjects with T1DM or T2DM.
* Must be able to read and sign the approved consent form.
* Registered into the LifeScan patient registry.
* Currently performing self monitoring of blood glucose ( SMBG)

Summary of Exclusion Criteria:

* Conflict of Interest - Prospective Participants will be excluded from enrollment if they are currently working for, have previously worked for, or have an immediate family member working for a company that manufactures or markets the type of products tested under the scope of this procedure.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of blood glucose ( BG) results between 3 LifeScan blood glucose monitoring systems ( BGMS). | Within 24 hours
  Comparison of Blood glucose results between 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus.) using capillary and Venous blood samples.
BG results of 3 BGMSs vs hospital's laboratory biochemistry analyser. | Within 24 hours
  Blood glucose result on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus.) compared to hospitals own laboratory biochemistry analyser using venous blood.
BG results of 3 BGMSs vs LifeScan reference instrument ( YSI 2300) | Within 24 hours
  Blood glucose result on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus.) compared to LifeScan's reference instrument ( YSI 2300) using venous and capillary blood.
Venous blood collected for impact assessment of Biochemistry parameters on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus). | Within 24 hours
  The following biochemistry parameters were analysed in mmol/l: Calcium, adjusted calcium, Chloride, Glucose, Potassium, Sodium, Triglycerides, urea, urate, Total Co2
Venous blood collected for impact assessment of Biochemistry parameters on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus). | Within 24 hours
  The following biochemistry parameters were analysed in Umol/l: creatine, Bilirubin, total bilirubin, direct bilirubin
Venous blood collected for impact assessment of Biochemistry parameters on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus). | Within 24 hours
  The following biochemistry parameters were analysed in U/L: ALT, ALK. Phos, LDH- Architect
Venous blood collected for impact assessment of Biochemistry parameters on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus). | Within 24 hours
  The following biochemistry parameters were analysed in G/L: Albumin, Total protein
Venous blood collected for impact assessment of Biochemistry parameters on 3 LifeScan Blood Glucose Monitoring Systems (OneTouch Ultra 2, OneTouch Verio, OneTouch SelectPlus). | Within 24 hours
  The following biochemistry parameters were analysed in (/1.73m2): eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Macleod, Study Director — LifeScan
Locations (3):
- United Kingdom (3):
  - Diabetes Centre, Heartlands Hospital, Birmingham
  - NHS Lothian, Edinburgh
  - Highland Diabetes Institute, Inverness

IPD SHARING:
Plan to Share IPD: No